CLINICAL TRIAL: NCT00312494
Title: A Three-Week, Double-Blind, Multicenter, Placebo-Controlled Study Evaluating the Efficacy and Safety of Add-On Oral Ziprasidone in Subjects With Acute Mania Treated With Lithium or Divalproex
Brief Title: 3-week Study to Evaluate Efficacy and Safety of Ziprasidone With Either Lithium or Divalproex in Acutely Manic Subjects
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: A1281143
Record Dates: First submitted 2006-04-06; First posted 2006-04-10 (Estimated); Results first posted 2010-01-22 (Estimated); Last update posted 2021-03-29 (Actual); Status verified 2021-03

CONDITIONS: Bipolar Disorder
MeSH Terms: conditions — Bipolar Disorder | interventions — ziprasidone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Ziprasidone 20-40mg twice a day (BID) (Experimental)
  Interventions: Drug: Ziprasidone
- Ziprasidone 60-80mg BID (Experimental)
  Interventions: Drug: Ziprasidone

INTERVENTIONS:
Drug: Placebo — Placebo with mood stabilizer (either lithium or divalproex)
  Arms: Placebo
Drug: Ziprasidone — Flexible dosing, 20-40mg BID, with a mood stabilizer (either lithium or divalproex)
  Other Names: Geodon, Zeldox
  Arms: Ziprasidone 20-40mg twice a day (BID)
Drug: Ziprasidone — Flexible dosing, 60-80mg BID, with a mood stabilizer (either lithium or divalproex)
  Other Names: Geodon, Zeldox
  Arms: Ziprasidone 60-80mg BID

SUMMARY:
3-week study to evaluate efficacy and safety of ziprasidone with either lithium or divalproex in acutely manic subjects

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have a primary diagnosis of Bipolar I Disorder, most recent episode manic (296.4x), or mixed (296.6x) as defined in Diagnostic and Statistical Manual of Mental Disorders - Text Revision (DSM-IV TR) and determined by the Mini International Neuropsychiatric Interview (MINI).
* At screening and at baseline (within 12 hours prior to the first dose of double-blind medication) subjects must have a Young Mania Rating Scale score of 18 or higher.
* Subjects must be actively receiving lithium or divalproex for their bipolar disorder in order to be considered for this study.

Exclusion Criteria:

* Subjects with a Diagnostic and Statistical Manual of Mental Disorders IV- Text Revision (DSM-IV TR) diagnosis of schizophrenia (295.XX), schizoaffective disorder (295.70), schizophreniform disorder (295.40), delusional disorder (297.1), or psychotic disorder not otherwise specified (NOS) (298.9).
* Subjects with other DSM-IV-TR Axis I or Axis II disorders (in addition to Bipolar I disorder) are ineligible if the comorbid condition is clinically unstable, requires treatment, or has been a primary focus of treatment within the 6-month period prior to screening.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 680 (Actual)
Dates: Start 2006-04; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (54):
- United States (54):
  - Pfizer Investigational Site, Dothan, Alabama
  - Pfizer Investigational Site, Scottsdale, Arizona
  - Pfizer Investigational Site, Little Rock, Arkansas
  - Pfizer Investigational Site, Cerritos, California
  - Pfizer Investigational Site, Costa Mesa, California
  - Pfizer Investigational Site, Escondido, California
  - Pfizer Investigational Site, Glendale, California
  - Pfizer Investigational Site, Huntington Beach, California
  - Pfizer Investigational Site, Los Angeles, California
  - Pfizer Investigational Site, National City, California
  - Pfizer Investigational Site, Oceanside, California
  - Pfizer Investigational Site, San Diego, California
  - Pfizer Investigational Site, Torrance, California
  - Pfizer Investigational Site, Hartford, Connecticut
  - Pfizer Investigational Site, New Britain, Connecticut
  - Pfizer Investigational Site, DeLand, Florida
  - Pfizer Investigational Site, Fort Lauderdale, Florida
  - Pfizer Investigational Site, Gainesville, Florida
  - Pfizer Investigational Site, Hollywood, Florida
  - Pfizer Investigational Site, Jacksonville, Florida
  - Pfizer Investigational Site, Lauderhill, Florida
  - Pfizer Investigational Site, North Miami, Florida
  - Pfizer Investigational Site, Atlanta, Georgia
  - Pfizer Investigational Site, Honolulu, Hawaii
  - Pfizer Investigational Site, Des Plaines, Illinois
  - Pfizer Investigational Site, Hoffman Estates, Illinois
  - Pfizer Investigational Site, Schaumburg, Illinois
  - Pfizer Investigational Site, Greenwood, Indiana
  - Pfizer Investigational Site, Prairie Village, Kansas
  - Pfizer Investigational Site, Glen Burnie, Maryland
  - Pfizer Investigational Site, Flowood, Mississippi
  - Pfizer Investigational Site, Kansas City, Missouri
  - Pfizer Investigational Site, Saint Charles, Missouri
  - Pfizer Investigational Site, St Louis, Missouri
  - Pfizer Investigational Site, Las Vegas, Nevada
  - Pfizer Investigational Site, Clementon, New Jersey
  - Pfizer Investigational Site, Princeton, New Jersey
  - Pfizer Investigational Site, Amityville, New York
  - Pfizer Investigational Site, Buffalo, New York
  - Pfizer Investigational Site, Cedarhurst, New York
  - Pfizer Investigational Site, Elmsford, New York
  - Pfizer Investigational Site, Raleigh, North Carolina
  - Pfizer Investigational Site, Cincinnati, Ohio
  - Pfizer Investigational Site, Cleveland, Ohio
  - Pfizer Investigational Site, Oklahoma City, Oklahoma
  - Pfizer Investigational Site, Philadelphia, Pennsylvania
  - Pfizer Investigational Site, Charleston, South Carolina
  - Pfizer Investigational Site, Dallas, Texas
  - Pfizer Investigational Site, Irving, Texas
  - Pfizer Investigational Site, Plano, Texas
  - Pfizer Investigational Site, San Antonio, Texas
  - Pfizer Investigational Site, Richmond, Virginia
  - Pfizer Investigational Site, Bellevue, Washington
  - Pfizer Investigational Site, Kirkland, Washington

REFERENCES:
- [Derived] Sachs GS, Vanderburg DG, Edman S, Karayal ON, Kolluri S, Bachinsky M, Cavus I. Adjunctive oral ziprasidone in patients with acute mania treated with lithium or divalproex, part 2: influence of protocol-specific eligibility criteria on signal detection. J Clin Psychiatry. 2012 Nov;73(11):1420-5. doi: 10.4088/JCP.11m07389. PMID 23218158
- [Derived] Sachs GS, Vanderburg DG, Karayal ON, Kolluri S, Bachinsky M, Cavus I. Adjunctive oral ziprasidone in patients with acute mania treated with lithium or divalproex, part 1: results of a randomized, double-blind, placebo-controlled trial. J Clin Psychiatry. 2012 Nov;73(11):1412-9. doi: 10.4088/JCP.11m07388. PMID 23218157
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A1281143&StudyName=3-week%20study%20to%20evaluate%20efficacy%20and%20safety%20of%20ziprasidone%20with%20either%20lithium%20or%20divalproex%20in%20acutely%20manic%20subjects

RESULTS

PARTICIPANT FLOW:
Groups:
- Ziprasidone (Higher Dose): Ziprasidone 120 to 160 mg daily + Mood Stabilizer
- Ziprasidone (Lower Dose): Ziprasidone 40 to 80 mg daily + Mood Stabilizer
- Placebo: Placebo (matching ziprasidone higher dose or ziprasidone lower dose) + Mood Stabilizer
Period: Overall Study
Arm/Group | Ziprasidone (Higher Dose) | Ziprasidone (Lower Dose) | Placebo
Started | 232 | 226 | 222
Received Study Treatment | 223 (1 subject randomized to higher dose; received lower dose at baseline, higher dose weeks 1 and 2.) | 216 | 217
Completed | 161 (1 subject randomized to higher dose; received lower dose baseline and/or week 1; higher dose week 2.) | 168 | 179
Not Completed | 71 | 58 | 43
Not completed — Randomized; not treated with study drug | 9 | 10 | 5
Not completed — Adverse Event | 33 | 15 | 11
Not completed — Lack of Efficacy | 4 | 6 | 8
Not completed — Laboratory abnormality | 1 | 0 | 0
Not completed — Lost to Follow-up | 8 | 8 | 8
Not completed — Withdrawal by Subject | 6 | 9 | 10
Not completed — Other | 10 | 10 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ziprasidone (Higher Dose) | Ziprasidone (Lower Dose) | Placebo | Total
Number analyzed (Participants) | 223 | 216 | 217 | 656
Age, Customized [Number; unit: participants]
  <18 years | 0 | 0 | 0 | 0
  Between 18 and 44 years | 125 | 124 | 126 | 375
  Between 45 and 64 years | 96 | 92 | 90 | 278
  >=65 years | 2 | 0 | 1 | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 100 | 108 | 110 | 318
  Male | 123 | 108 | 107 | 338

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Week 3 in Young Mania Rating Scale (YMRS)
Description: YMRS is an 11-item scale (elevated mood, increased motor activity-energy, sexual interest, sleep, irritability, speech [rate and amount], language-thought disorder, content, disruptive-aggressive behavior, appearance, and insight) used to assess the severity of manic symptoms and effect of treatment on mania severity. Seven items ranked on scale from 0 to 4; 4 items ranked 0 to 8. Total possible score 0 to 60: higher scores indicate greater severity. Change calculated as mean of (value of YMRS score at observation minus baseline value).
Time Frame: Baseline, Week 3
Population: Intent to Treat population (ITT): all randomized subjects who received at least 1 dose of double-blind medication, who had 1 baseline and at least 1 post-baseline primary efficacy evaluation; excluding data from 2 sites that were closed due to Good Clinical Practices (GCP) deviations.
Measure: Least Squares Mean (Standard Error); unit: scores on scale
Arm/Group | Ziprasidone (Higher Dose) | Ziprasidone (Lower Dose) | Placebo
Number analyzed (Participants) | 211 | 210 | 201
scores on scale | -10.19 (0.78) | -10.95 (0.80) | -9.47 (0.83)
Statistical Analysis 1: Comparison: Ziprasidone (Lower Dose) vs Placebo; N=135/arm (405 total) for 85% power for 2-sample t-test (2-sided alpha=0.05) based on true mean difference=3.5 and SD=10. Interim Analysis (IA) to validate sample-size assumptions and adjust sample-size if needed. Based on IA results total sample-size increased to N=223/arm (669 total) to maintain desired power. Null Hypothesis=No statistically significant difference between add-on ziprasidone (higher, lower dose) and add-on placebo groups with respect to the population mean for primary endpoint; Test type: Superiority or Other; p = 0.1077, Mixed Models Analysis — The p-values reported are unadjusted for multiple comparisons. Dunnet's procedure for multiple dose comparisons to placebo was used for primary efficacy measure at Week 3
Statistical Analysis 2: Comparison: Ziprasidone (Higher Dose) vs Placebo; Week 3 Mixed Model Repeated Measures (MMRM) with model terms: treatment, length of prior lithium/divalproex usage, type of mood stabilizer therapy, rapid cycling, hospitalization status, visit, treatment by visit interaction, and baseline YMRS total score. Tests were 2-sided and performed at the 0.05 significance level; Test type: Superiority or Other; p = 0.4274, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]

2. Secondary Outcome: Change From Baseline to Week 1 and Week 2 in YMRS
Description: as for outcome 1
Time Frame: Baseline, Week 1, Week 2
Population: ITT population excluding data from 2 sites that were closed to GCP deviations; (n)=number of subjects for ziprasidone (higher dose), ziprasidone (lower dose), and placebo, respectively.
Measure: Least Squares Mean (Standard Error); unit: scores on scale
Arm/Group | Ziprasidone (Higher Dose) | Ziprasidone (Lower Dose) | Placebo
Number analyzed (Participants) | 211 | 210 | 201
scores on scale
  Week 1 (n=202, 205, 200) | -4.38 (0.65) | -4.56 (0.65) | -5.10 (0.70)
  Week 2 (n=178, 188, 186) | -7.10 (0.72) | -7.56 (0.73) | -8.24 (0.76)
Statistical Analysis 1: Comparison: Ziprasidone (Lower Dose) vs Placebo; Week 1 MMRM with model terms: treatment, length of prior lithium/divalproex usage, type of mood stabilizer therapy, rapid cycling, hospitalization status, visit, treatment by visit interaction, and baseline YMRS total score; Test type: Superiority or Other; p = 0.4025, Mixed Models Analysis — The p-values reported are unadjusted for multiple comparisons
Statistical Analysis 2: Comparison: Ziprasidone (Higher Dose) vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.2830, Mixed Models Analysis — The p-values reported are unadjusted for multiple comparisons
Statistical Analysis 3: Comparison: Ziprasidone (Lower Dose) vs Placebo; Week 2 MMRM with model terms: treatment, length of prior lithium/divalproex usage, type of mood stabilizer therapy, rapid cycling, hospitalization status, visit, treatment by visit interaction, and baseline YMRS total score; Test type: Superiority or Other; p = 0.4125, Mixed Models Analysis — The p-values reported are unadjusted for multiple comparisons
Statistical Analysis 4: Comparison: Ziprasidone (Higher Dose) vs Placebo; [analysis description as in outcome 2, analysis 3]; Test type: Superiority or Other; p = 0.1527, Mixed Models Analysis — The p-values reported are unadjusted for multiple comparisons

3. Secondary Outcome: Change From Baseline in Montgomery Asberg Depression Rating Scale (MADRS) Total Scores
Description: MADRS is a 10-item clinician rated scale to measure overall severity of depressive symptoms (apparent sadness, reported sadness, inner tension, reduced sleep, reduced appetite, concentration difficulties, lassitude, inability to feel, pessimistic thoughts, suicidal thoughts); rated on a 7-point Likert scale 0 (normal) to 6 (most abnormal) with anchors at 2-point intervals; total score 0 to 44 (higher score indicates greater severity of symptoms). Change calculated as mean of (value of MADRS score at observation minus baseline value).
Time Frame: Baseline, Week 1, Week 2, Week 3
Population: ITT population excluding data from 2 sites that were closed due to GCP deviations; (n)=number of subjects for ziprasidone (higher dose), ziprasidone (lower dose), and placebo, respectively.
Measure: Least Squares Mean (Standard Error); unit: scores on scale
Arm/Group | Ziprasidone (Higher Dose) | Ziprasidone (Lower Dose) | Placebo
Number analyzed (Participants) | 211 | 210 | 201
scores on scale
  Week 1 (n=202, 205, 200) | -2.16 (0.52) | -2.47 (0.49) | -1.11 (0.63)
  Week 2 (n=178, 188, 186) | -3.27 (0.57) | -3.24 (0.55) | -1.71 (0.66)
  Week 3 (n=163, 172, 170) | -4.20 (0.63) | -3.79 (0.64) | -2.90 (0.70)
Statistical Analysis 1: Comparison: Ziprasidone (Lower Dose) vs Placebo; Week 1 MMRM with model terms: treatment, length of prior lithium/divalproex usage, type of mood stabilizer therapy, rapid cycling, hospitalization status, visit, treatment by visit interaction, and baseline MADRS total score; Test type: Superiority or Other; p = 0.0101, Mixed Models Analysis — The p-values reported are unadjusted for multiple comparisons
Statistical Analysis 2: Comparison: Ziprasidone (Higher Dose) vs Placebo; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.0694, Mixed Models Analysis — The p-values reported are unadjusted for multiple comparisons
Statistical Analysis 3: Comparison: Ziprasidone (Lower Dose) vs Placebo; Week 2 MMRM with model terms: treatment, length of prior lithium/divalproex usage, type of mood stabilizer therapy, rapid cycling, hospitalization status, visit, treatment by visit interaction, and baseline MADRS total score; Test type: Superiority or Other; p = 0.0183, Mixed Models Analysis — The p-values reported are unadjusted for multiple comparisons
Statistical Analysis 4: Comparison: Ziprasidone (Higher Dose) vs Placebo; [analysis description as in outcome 3, analysis 3]; Test type: Superiority or Other; p = 0.0176, Mixed Models Analysis — The p-values reported are unadjusted for multiple comparisons
Statistical Analysis 5: Comparison: Ziprasidone (Lower Dose) vs Placebo; Week 3 MMRM with model terms: treatment, length of prior lithium/divalproex usage, type of mood stabilizer therapy, rapid cycling, hospitalization status, visit, treatment by visit interaction, and baseline MADRS total score; Test type: Superiority or Other; p = 0.2302, Mixed Models Analysis — The p-values reported are unadjusted for multiple comparisons
Statistical Analysis 6: Comparison: Ziprasidone (Higher Dose) vs Placebo; [analysis description as in outcome 3, analysis 5]; Test type: Superiority or Other; p = 0.0796, Mixed Models Analysis — The p-values reported are unadjusted for multiple comparisons

4. Secondary Outcome: Change From Baseline in Clinical Global Impression Scale - Severity (CGI-S) Score
Description: CGI-S is a single-item clinician rated scale used to assess global severity of bipolar illness based on an overall evaluation of symptoms of bipolar mania, associated behavioral symptoms, and condition of the subject. Rating ranges from 1 (normal, not at all ill) to 7 (among the most severely ill subjects); higher score = more affected. Change calculated as mean of (value of CGI-S score at observation minus baseline value).
Time Frame: Baseline, Week 1, Week 2, Week 3
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: scores on scale
Arm/Group | Ziprasidone (Higher Dose) | Ziprasidone (Lower Dose) | Placebo
Number analyzed (Participants) | 211 | 210 | 201
scores on scale
  Week 1 (n=202, 206, 200) | -0.35 (0.06) | -0.43 (0.06) | -0.39 (0.07)
  Week 2 (n=178, 188, 186) | -0.70 (0.08) | -0.74 (0.07) | -0.73 (0.09)
  Week 3 (n=163, 172, 171) | -0.94 (0.08) | -1.13 (0.09) | -1.00 (0.09)
Statistical Analysis 1: Comparison: Ziprasidone (Lower Dose) vs Placebo; Week 1 MMRM with model terms: treatment, length of prior lithium/divalproex usage, type of mood stabilizer therapy, rapid cycling, hospitalization status, visit, treatment by visit interaction, and baseline as covariate; Test type: Superiority or Other; p = 0.6191, Mixed Models Analysis — The p-values reported are unadjusted for multiple comparisons
Statistical Analysis 2: Comparison: Ziprasidone (Higher Dose) vs Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.5629, Mixed Models Analysis — The p-values reported are unadjusted for multiple comparisons
Statistical Analysis 3: Comparison: Ziprasidone (Lower Dose) vs Placebo; Week 2 MMRM with model terms: treatment, length of prior lithium/divalproex usage, type of mood stabilizer therapy, rapid cycling, hospitalization status, visit, treatment by visit interaction, and baseline as covariate; Test type: Superiority or Other; p = 0.9049, Mixed Models Analysis — The p-values reported are unadjusted for multiple comparisons
Statistical Analysis 4: Comparison: Ziprasidone (Higher Dose) vs Placebo; [analysis description as in outcome 4, analysis 3]; Test type: Superiority or Other; p = 0.7153, Mixed Models Analysis — The p-values reported are unadjusted for multiple comparisons
Statistical Analysis 5: Comparison: Ziprasidone (Lower Dose) vs Placebo; Week 3 MMRM with model terms: treatment, length of prior lithium/divalproex usage, type of mood stabilizer therapy, rapid cycling, hospitalization status, visit, treatment by visit interaction, and baseline as covariate; Test type: Superiority or Other; p = 0.2420, Mixed Models Analysis — The p-values reported are unadjusted for multiple comparisons
Statistical Analysis 6: Comparison: Ziprasidone (Higher Dose) vs Placebo; [analysis description as in outcome 4, analysis 5]; Test type: Superiority or Other; p = 0.6121, Mixed Models Analysis — The p-values reported are unadjusted for multiple comparisons

5. Secondary Outcome: Clinical Global Impression - Improvement (CGI-I) Scale Scores
Description: CGI-I is a single-item clinician rated scale used to assess global improvement in the subject's clinical state (bipolar mania) in response to study treatment and as compared to their status at pre-treatment baseline. Scores range from 1 (very much improved) to 4 (no change) to 7 (very much worse); higher score = more affected.
Time Frame: Week 1, Week 2, Week 3
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: scores on scale
Arm/Group | Ziprasidone (Higher Dose) | Ziprasidone (Lower Dose) | Placebo
Number analyzed (Participants) | 211 | 210 | 201
scores on scale
  Week 1 (n=202, 206, 200) | 3.34 (0.09) | 3.34 (0.09) | 3.38 (0.08)
  Week 2 (n=178, 188, 186) | 3.02 (0.10) | 2.91 (0.09) | 2.98 (0.10)
  Week 3 (n=163, 172, 171) | 2.65 (0.11) | 2.57 (0.11) | 2.72 (0.11)
Statistical Analysis 1: Comparison: Ziprasidone (Lower Dose) vs Placebo; Week 1 MMRM with model terms: treatment, length of prior lithium/divalproex usage, type of mood stabilizer therapy, rapid cycling, hospitalization status, visit, and treatment by visit interaction; Test type: Superiority or Other; p = 0.6138, Mixed Models Analysis — The p-values reported are unadjusted for multiple comparisons
Statistical Analysis 2: Comparison: Ziprasidone (Higher Dose) vs Placebo; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p = 0.6536, Mixed Models Analysis — The p-values reported are unadjusted for multiple comparisons
Statistical Analysis 3: Comparison: Ziprasidone (Lower Dose) vs Placebo; Week 2 MMRM with model terms: treatment, length of prior lithium/divalproex usage, type of mood stabilizer therapy, rapid cycling, hospitalization status, visit, and treatment by visit interaction; Test type: Superiority or Other; p = 0.4758, Mixed Models Analysis — The p-values reported are unadjusted for multiple comparisons
Statistical Analysis 4: Comparison: Ziprasidone (Higher Dose) vs Placebo; [analysis description as in outcome 5, analysis 3]; Test type: Superiority or Other; p = 0.7581, Mixed Models Analysis — The p-values reported are unadjusted for multiple comparisons
Statistical Analysis 5: Comparison: Ziprasidone (Lower Dose) vs Placebo; Week 3 MMRM with model terms: treatment, length of prior lithium/divalproex usage, type of mood stabilizer therapy, rapid cycling, hospitalization status, visit, and treatment by visit interaction; Test type: Superiority or Other; p = 0.2221, Mixed Models Analysis — The p-values reported are unadjusted for multiple comparisons
Statistical Analysis 6: Comparison: Ziprasidone (Higher Dose) vs Placebo; [analysis description as in outcome 5, analysis 5]; Test type: Superiority or Other; p = 0.5665, Mixed Models Analysis — The p-values reported are unadjusted for multiple comparisons

6. Secondary Outcome: Change From Baseline in Positive and Negative Syndrome Scale (PANSS) Score
Description: PANSS is a 30-item scale to measure severity of psychopathology (16 items); positive scale (7 items); negative scale (7 items); summarized as positive score, negative score, and total score. Scores rated 1 (absent symptoms) to 7 (extreme); total score range 30 to 210: higher score indicates greater severity. Change calculated as mean of (value of PANSS score at observation minus baseline value).
Time Frame: Baseline, Week 3
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: scores on scale
Arm/Group | Ziprasidone (Higher Dose) | Ziprasidone (Lower Dose) | Placebo
Number analyzed (Participants) | 211 | 210 | 201
scores on scale
  Week 3 total score (n=198, 199, 189) | -4.87 (1.86) | -5.34 (1.68) | -3.44 (1.84)
  Week 3 positive score (n=198, 199, 189) | -1.94 (0.52) | -2.26 (0.52) | -1.56 (0.56)
  Week 3 negative score (n=198, 199, 189) | -0.58 (0.51) | -0.43 (0.51) | -0.20 (0.52)
Statistical Analysis 1: Comparison: Ziprasidone (Lower Dose) vs Placebo; Week 3 total score MMRM with model terms: treatment, length of prior lithium/divalproex usage, type of mood stabilizer therapy, rapid cycling, hospitalization status, visit, treatment by visit interaction, and baseline PANSS total score; Test type: Superiority or Other; p = 0.1063, Mixed Models Analysis — The p-values reported are unadjusted for multiple comparisons
Statistical Analysis 2: Comparison: Ziprasidone (Higher Dose) vs Placebo; [analysis description as in outcome 6, analysis 1]; Test type: Superiority or Other; p = 0.2499, Mixed Models Analysis — The p-values reported are unadjusted for multiple comparisons
Statistical Analysis 3: Comparison: Ziprasidone (Lower Dose) vs Placebo; Week 3 positive score MMRM with model terms: treatment, length of prior lithium/divalproex usage, type of mood stabilizer therapy, rapid cycling, hospitalization status, visit, treatment by visit interaction, and baseline PANSS positive score; Test type: Superiority or Other; p = 0.0876, Mixed Models Analysis — The p-values reported are unadjusted for multiple comparisons
Statistical Analysis 4: Comparison: Ziprasidone (Higher Dose) vs Placebo; [analysis description as in outcome 6, analysis 3]; Test type: Superiority or Other; p = 0.3623, Mixed Models Analysis — The p-values reported are unadjusted for multiple comparisons
Statistical Analysis 5: Comparison: Ziprasidone (Lower Dose) vs Placebo; Week 3 negative score MMRM with model terms: treatment, length of prior lithium/divalproex usage, type of mood stabilizer therapy, rapid cycling, hospitalization status, visit, treatment by visit interaction, and baseline PANSS negative score; Test type: Superiority or Other; p = 0.4686, Mixed Models Analysis — The p-values reported are unadjusted for multiple comparisons
Statistical Analysis 6: Comparison: Ziprasidone (Higher Dose) vs Placebo; [analysis description as in outcome 6, analysis 5]; Test type: Superiority or Other; p = 0.2202, Mixed Models Analysis — The p-values reported are unadjusted for multiple comparisons

7. Secondary Outcome: Change From Baseline in Global Assessment of Functioning (GAF) Score
Description: GAF measures the severity of illness-related impairment in psychological, social, and occupational functioning; rated on a 100-point scale (single score of 1 to 100) with 100 indicating superior functioning. Change calculated as mean of (value of GAF score at observation minus baseline value).
Time Frame: Baseline, Week 3
Population: ITT population excluding data from 2 sites that were closed due to GCP deviations.
Measure: Least Squares Mean (Standard Error); unit: scores on scale
Arm/Group | Ziprasidone (Higher Dose) | Ziprasidone (Lower Dose) | Placebo
Number analyzed (Participants) | 211 | 210 | 201
scores on scale | 8.79 (1.23) | 9.62 (1.25) | 7.79 (1.22)
Statistical Analysis 1: Comparison: Ziprasidone (Lower Dose) vs Placebo; Week 3 MMRM with model terms: treatment, length of prior lithium/divalproex usage, type of mood stabilizer therapy, rapid cycling, hospitalization status, visit, treatment by visit interaction, and baseline GAF score; Test type: Superiority or Other; p = 0.0728, Mixed Models Analysis — The p-values reported are unadjusted for multiple comparisons
Statistical Analysis 2: Comparison: Ziprasidone (Higher Dose) vs Placebo; [analysis description as in outcome 7, analysis 1]; Test type: Superiority or Other; p = 0.3174, Mixed Models Analysis — The p-values reported are unadjusted for multiple comparisons

8. Secondary Outcome: Change From Baseline in Longitudinal Interval Follow-up Evaluation Range of Impaired Functioning (LIFE-RIFT) Score
Description: LIFE-RIFT measures severity of illness-related impairment in 4 domains: work, interpersonal relations, recreation, and global satisfaction; has a total score and individual domain scores. Domain scores range from 1 to 5 (scores ≥ 2 reflect impaired functioning). Total score is sum of the 4 domains with range of 4 (very good) to 20 (very poor): higher scores indicate greater impairment. Change calculated as mean of (value of LIFE-RIFT score at observation minus baseline value).
Time Frame: Baseline, Week 3
Population: ITT population excluding data from 2 sites that were closed due to GCP deviations.
Measure: Least Squares Mean (Standard Error); unit: scores on scale
Arm/Group | Ziprasidone (Higher Dose) | Ziprasidone (Lower Dose) | Placebo
Number analyzed (Participants) | 211 | 210 | 201
scores on scale | -1.68 (0.45) | -1.58 (0.50) | -1.27 (0.46)
Statistical Analysis 1: Comparison: Ziprasidone (Lower Dose) vs Placebo; Week 3 MMRM with model terms: treatment, length of prior lithium/divalproex usage, type of mood stabilizer therapy, rapid cycling, hospitalization status, visit, treatment by visit interaction, and baseline LIFE-RIFT total score; Test type: Superiority or Other; p = 0.4460, Mixed Models Analysis — The p-values reported are unadjusted for multiple comparisons
Statistical Analysis 2: Comparison: Ziprasidone (Higher Dose) vs Placebo; [analysis description as in outcome 8, analysis 1]; Test type: Superiority or Other; p = 0.3253, Mixed Models Analysis — The p-values reported are unadjusted for multiple comparisons

9. Secondary Outcome: Anonymized Pharmacogenomic Blood Draw
Description: Anonymized pharmacogenomic blood draw to evaluate the pharmacogenomic basis for ziprasidone treatment responsivity.
Time Frame: Baseline
Population: All subjects eligible (optional consent); samples were not to be analyzed as part of the current protocol and the analysis was not to be covered by the statistical analysis plan.
Arm/Group | Ziprasidone (Higher Dose) | Ziprasidone (Lower Dose) | Placebo
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Description: Safety population: all randomized subjects who were administered at least 1 dose of double-blind medication; includes data from the 2 sites that were closed due to GCP deviations.
Arm/Group | Ziprasidone (Higher Dose) | Ziprasidone (Lower Dose) | Placebo
Serious Adverse Events (participants affected / at risk) | 5/223 | 4/216 | 4/217
Other Adverse Events (participants affected / at risk) | 134/223 | 99/216 | 82/217
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ziprasidone (Higher Dose) (N=223) | Ziprasidone (Lower Dose) (N=216) | Placebo (N=217)
Chest pain (General disorders) | 0 | 0 | 1
Cellulitis (Infections and infestations) | 1 | 0 | 0
Intentional overdose (Injury, poisoning and procedural complications) | 0 | 1 | 0
Overdose (Injury, poisoning and procedural complications) | 0 | 1 | 1
Thermal burn (Injury, poisoning and procedural complications) | 1 | 0 | 0
Blood pressure increased (Investigations) | 0 | 1 | 0
Anterograde amnesia (Nervous system disorders) | 0 | 1 | 0
Acute psychosis (Psychiatric disorders) | 1 | 0 | 0
Agitation (Psychiatric disorders) | 1 | 0 | 0
Alcohol abuse (Psychiatric disorders) | 0 | 1 | 0
Bipolar I disorder (Psychiatric disorders) | 1 | 1 | 1
Drug abuse (Psychiatric disorders) | 0 | 1 | 0
Emotional disorder (Psychiatric disorders) | 0 | 0 | 1
Suicide attempt (Psychiatric disorders) | 0 | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ziprasidone (Higher Dose) (N=223) | Ziprasidone (Lower Dose) (N=216) | Placebo (N=217)
Abdominal discomfort (Gastrointestinal disorders) | 6 | 2 | 2
Diarrhoea (Gastrointestinal disorders) | 12 | 10 | 7
Dry mouth (Gastrointestinal disorders) | 6 | 1 | 3
Nausea (Gastrointestinal disorders) | 11 | 11 | 13
Salivary hypersecretion (Gastrointestinal disorders) | 5 | 4 | 0
Vomiting (Gastrointestinal disorders) | 13 | 6 | 4
Fatigue (General disorders) | 11 | 3 | 5
Nasopharyngitis (Infections and infestations) | 7 | 1 | 4
Upper respiratory tract infection (Infections and infestations) | 5 | 7 | 5
Increased appetite (Metabolism and nutrition disorders) | 1 | 5 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 5 | 1
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 4 | 6 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 | 7 | 2
Akathisia (Nervous system disorders) | 15 | 8 | 5
Dizziness (Nervous system disorders) | 16 | 5 | 6
Extrapyramidal disorder (Nervous system disorders) | 11 | 4 | 1
Headache (Nervous system disorders) | 10 | 19 | 16
Sedation (Nervous system disorders) | 33 | 17 | 18
Somnolence (Nervous system disorders) | 26 | 19 | 5
Tremor (Nervous system disorders) | 12 | 6 | 7
Agitation (Psychiatric disorders) | 6 | 4 | 1
Anxiety (Psychiatric disorders) | 5 | 2 | 2
Insomnia (Psychiatric disorders) | 8 | 3 | 5
Restlessness (Nervous system disorders) | 6 | 3 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 5 | 1 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of < 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), < 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.